CLINICAL TRIAL: NCT06799169
Title: Management of Acute Tinnitus With Migraine Medications: A Randomized Clinical Trial
Brief Title: Management of Acute Tinnitus With Migraine Medications
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mehdi Abouzari, MD, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4863
Record Dates: First submitted 2024-08-29; First posted 2025-01-29 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-08

CONDITIONS: Tinnitus
Keywords: Tinnitus; Acute tinnitus; Atypical migraine; ringing in ears
MeSH Terms: conditions — Tinnitus; Migraine without Aura | interventions — Nortriptyline; Topiramate; Paroxetine; Verapamil

STUDY DESIGN:
Intervention Model Description: This study is an 8-week, randomized, double-blind, single-center clinical trial, consisting of two arms: Group N-T, a nortriptyline (7.5mg) plus topiramate (10mg) group and group V-P, a verapamil (30mg) plus paroxetine (4mg) group. Both groups may involve dose escalation from the initial dosage during the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The principal investigator, provider, lead researchers and the subjects will be masked throughout the duration of the clinical trial. Solely the clinical coordinator will be unmasked during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group N-T (Active Comparator): Nortriptyline (starting dose 7.5 mg) plus Topiramate (starting dose 10 mg) with appropriate dosage increase as necessary.
  The reported symptoms will dictate dosage adjustments. If symptoms do not improve, patients will be advised to increase their dosage by adding one additional pill, which equals an increase of nortriptyline by 7.5 mg and topiramate by 10 mg for one week until the next phone check-in. This process will continue until the patient reaches a maximum of 60mg for nortriptyline plus 80mg for topiramate for the duration of the 8 weeks (a total of 8 pills of each combination).
  Interventions: Drug: Nortriptyline; Drug: Topiramate
- Group V-P (Active Comparator): Verapamil (starting dose 30 mg) plus Paroxetine (starting dose 4 mg) with appropriate dosage increase as necessary.
  The reported symptoms will dictate dosage adjustments. If symptoms do not improve, patients will be advised to increase their dosage by adding one additional pill, which equals an increase of verapamil by 30 mg and paroxetine by 4 mg, for one week until the next phone check-in. This process will continue until the patient reaches a maximum of 240mg of verapamil plus 32mg of paroxetine for the duration of the 8 weeks (a total of 8 pills of each combination).
  Interventions: Drug: Paroxetine; Drug: Verapamil

INTERVENTIONS:
Drug: Nortriptyline — Nortriptyline (7.5 mg) plus Topiramate (10 mg) taken by mouth daily with appropriate dosage increase as necessary
  Other Names: Pamelor
  Arms: Group N-T
Drug: Topiramate — Nortriptyline (7.5 mg) plus Topiramate (10 mg) taken by mouth daily with appropriate dosage increase as necessary
  Other Names: Topamax
  Arms: Group N-T
Drug: Paroxetine — Verapamil (30 mg) plus Paroxetine (4 mg) taken by mouth daily with appropriate dosage increase as necessary
  Other Names: Paxil
  Arms: Group V-P
Drug: Verapamil — Verapamil (30 mg) plus Paroxetine (4 mg) taken by mouth daily with appropriate dosage increase as necessary
  Other Names: Calan SR
  Arms: Group V-P

SUMMARY:
Tinnitus represents one of the most common and distressing otologic problems, and it causes various somatic and psychological disorders that interfere with the quality of life. Despite too many research projects on finding the mechanism of tinnitus, its pathophysiology remains poorly understood. It is well understood that many factors, such as poor education, lower income, or occupational, and recreational activity associated with high noise exposure, influence the prevalence and risk of tinnitus. Although the economic and emotional impact of tinnitus is large, there is currently no FDA-approved medication to treat this condition. However, there are pharmacological options to address the stress, anxiety, and depression that are caused by tinnitus. In this project, the investigators intend to use medications for patients with acute tinnitus to decrease the impact of tinnitus in their daily lives and activities. There are some studies on medications treating tinnitus; however, there are few randomized clinical trials to prove the efficacy of the treatment. The frequency and loudness of tinnitus will be measured before and after the course. Functional MRI of the brain will be obtained to view any changes that may occur before and after the treatment.

DETAILED DESCRIPTION:
This study is 8-weeks in duration. There are two arms in the experiment: the first is nortriptyline (7.5 mg) plus topiramate (10 mg), the second is verapamil (240 mg) plus paroxetine (32 mg). This is a double-blinded trial. Participants will be randomized to one arm for the duration of the trial using simple randomization with a computer-generated number. Both groups may receive dosage increases weekly if symptoms do not improve. Symptomatic survey scores from each arm will be obtained before and after treatment and weekly. An unblinded clinical researcher will also become involved with patients' treatments as they start to report changes in symptoms in order to monitor their safety and provide advice on change in dosage if patients have questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate tinnitus.
* Male or female between the ages of 25 to 85 years.
* Subjects must be compliant with the medication and attend study visits.
* Must be able to read and write in the English language to provide consent.

Exclusion Criteria:

* Pregnancy will result in automatic exclusion from the study. Rule out of pregnancy will be done by urine pregnancy test to confirm the situation for all women who are of childbearing potential.
* Subjects with a history of an adverse reaction to medication being prescribed.
* Subjects suffering from a medical condition or have a history that may be concerning to the investigator's clinical opinion.
* All contraindications for the medications that prevent subjects from randomization will be considered as exclusion criteria.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index | 8 weeks
  The primary outcome endpoint is a Tinnitus Functional Index (TFI) score which comprehensively evaluates the negative impact of tinnitus across 8 domains each focusing on specific dimensions: Intrusive, Sense of control, Cognitive, Sleep, Auditory, Relaxation, Quality of life, and Emotional. The overall score ranges from 0 to 100. Changes 13 points in TFI are the Minimal Clinically Important Difference (MCID). Subjective improvement from baseline in tinnitus symptoms as measured by Tinnitus Functional Index (TFI). The TFI is scored from 0% to 100%, with higher scores indicating a more negative impact of tinnitus.

SECONDARY OUTCOMES:
Tinnitus Functional Index (TFI) | 8 weeks
  Subjective improvement from baseline in tinnitus symptoms as measured by Tinnitus Functional Index (TFI). The TFI is scored from 0% to 100%, with higher scores indicating a more negative impact of tinnitus.
Perceived Stress Scale (PSS) | 8 weeks
  Perceived Stress Scale (PSS) [Time Frame: 8 weeks] Subjective improvement in stress based on perceived stress scale (PSS). The PSS is scored from 0 to 40, with higher scores indicating higher perceived stress.
Patient Health Questionnaire (PHQ-9) | 8 weeks
  Subjective improvement in depression symptoms based on patient health questionnaire (PHQ). The PHQ is scored from 0 to 27, with a higher score indicating increased depression severity.
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  Subjective improvement in sleep quality based on sleep quality index (PSQI). The PSQI is scored from 0 to 21, with higher scores indicating worse quality of sleep.
Generalized Anxiety Disorder (GAD-7) | 8 weeks
  Subjective improvement in generalized anxiety based on general anxiety disorder (GAD-7). The GAD-7 is scored from 0 to 21, with higher scores indicating increased anxiety severity.
Visual Analog Scale (VAS) | 8 weeks
  Subjective improvement in tinnitus loudness severity based on a visual analog scale (VAS). The VAS is scored from 0 to 10, with a higher score representing an increased severity of tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Abouzari, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center ENT Clinic (Pavilion 2), Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
Final study results will not be shared with subjects. Upon the final appointment patient will be told of which medication they have been given. It will not be necessary to share the final results since the patient will know if their symptoms have improved- no lab value can be given to measure this. Since this study will be listed on clinicaltrials.gov, the overall study results will be available through that platform after the completion of the study.